CLINICAL TRIAL: NCT06061276
Title: Sequential bTAE-HAIC Combined With Lenvatinib and Camrelizumab for Intermediate-advanced Huge Hepatocellular Carcinoma
Brief Title: bTAE-HAIC Combined With System Therapy for Intermediate-advanced Huge HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Liver Project 3
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Liver Diseases; Hepatocellular Carcinoma; Immunotherapy; Camrelizumab; Lenvatinib
MeSH Terms: conditions — Liver Diseases; Carcinoma, Hepatocellular | interventions — lenvatinib; camrelizumab; Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bTAE-HAIC combined with Lenvatinib and Camrelizumab (Experimental): bTAE procedure was a 2.8-F microcatheter was super-selectively inserted into the tumor feeding artery using the coaxial technique. Then blank microspheres were used according to the tumor blood supply vessels (40-120um, 100-300um, 300-500um, 500-700um). Hepatic arterial infusion of oxaliplatin, fluorouracil, and leucovorin every 4 weeks.
  Interventions: Procedure: bTAE-HAIC; Drug: Lenvatinib; Drug: Camrelizumab

INTERVENTIONS:
Procedure: bTAE-HAIC — bTAE procedure was a 2.8-F microcatheter was superselectively inserted into the tumor feeding artery using the coaxial technique. Then blank microspheres were used according to the tumor blood supply vessels (40-120um, 100-300um, 300-500um, 500-700um). The microcatheter was reserved at the proper/left/right hepatic artery according tumor location. After the patient returned to the ward, the following FOLFOX-based regime was intra-arterially administered through the microcatheter. The FOLFOX regimen was administered via the hepatic artery as follows: 85 or 135 mg/m2 oxaliplatin from hour 0 to 2 on day 1, and 400 mg/m2 leucovorin from hour 2 to 4 on day 1, and 400 mg/m2 fluorouracil bolus at hour 5 on the day 1; and 2400 mg/m2 fluorouracil over 46 h on days 1 and 2.
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.
  Other Names: TKI inhibits
Drug: Camrelizumab — 200mg intravenously every 2 weeks
  Other Names: programmed cell death protein-1 (PD-1) antibody

SUMMARY:
This study intends to evaluate the efficacy and safety of blank- microsphere transcatheter arterial embolization-hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin (bTAE-HAIC) plus Lenvatinib and Camrelizumab for patients with intermediate-advanced huge hepatocellular carcinoma.

DETAILED DESCRIPTION:
Blank-microsphere transcatheter arterial embolization (bTAE) and hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin are effective and safe for hepatocellular carcinoma. Lenvatinib is non-inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma. Camrelizumab, a programmed cell death protein-1 (PD-1) inhibitor, is effective and tolerable in patients with unresectable hepatocellular carcinoma. No study has evaluated bTAE-HAIC plus Lenvatinib and Camrelizumab. Thus, the investigators carried out this prospective, single-arm study to find out it.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of HCC.
2. Age between 18 and 75 years;
3. The maximum tumor size ≥10 cm, and the total tumor size ≥15 cm;
4. Intermediate-advanced huge HCC, advanced HCC with PVTT type I or type II or limited metastases (≤5).
5. Child-Pugh class A or B;
6. Eastern Cooperative Group performance status (ECOG) score of 0-2;
7. Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3
8. Prothrombin time ≤18s or international normalized ratio < 1.7.
9. Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

1. Diffuse HCC;
2. Extrahepatic metastasis >5;
3. Obstructive PVTT involving the main portal vein.
4. Serious medical comorbidities.
5. Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
6. Known history of HIV
7. History of organ allograft
8. Known or suspected allergy to the investigational agents or any agent given in association with this trial.
9. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
10. Evidence of bleeding diathesis.
11. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as

SECONDARY OUTCOMES:
Progression free survival (PFS) | 6 months
  PFS is defined as the time from the date of inclusion to the date of the first objectively documented tumor progression or death due to any cause.

OTHER OUTCOMES:
Overall survival (OS) | 12 months
  OS is the length of time from the date of inclusion until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimei Hunag, MD, Study Director — Sun Yat-sen University; Jinhua Huang, Profession, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No